CLINICAL TRIAL: NCT00835809
Title: Multi Marker Approach Interest in Emergency in Acute Respiratory Insufficiency Diagnostic
Acronym: BIO-IRA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Regional Clinical Research (Other)
Responsible Party: Ms Claire ARA SOMOHANO, Service de réanimation médicale
Other Study IDs: 0811; 2008-A00703-52 (Registry Identifier: ID RCB)
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Acute Respiratory Insufficiency
Keywords: Acute respiratory insufficiency respiratory; Biomarkers; Emergency; Intensive care unit; Prospective; Patient hospitalize in emergency or in intensive care unit; for acute respiratory insufficiency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Protein sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute respiratory diseases.: Patient admit in emergency or intensive care unite with acute respiratory insufficiency.

SUMMARY:
Biomarkers have an interest in clinic diagnostic ,therapeutic and prognosis in pathophysiologic situation including cardiovascular.But interest of biomarkers in diagnostic care of severe acute respiratory insufficiency remains to clear.

We propose to determine the more relevant marker combination in this case.

DETAILED DESCRIPTION:
In urgence of a severe acute respiratory insufficiency,for thanks to an approach diagnostic, therapeutic and prognostic we propose to determine the more relevant biomarker combination.

An expert committee will compare the biomarker diagnostic and prognostic relevance thanks to all elements clinico-biological and patient monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Oxygen saturation below or equal to 92% in ambient air.
* Respiratory frequence above 25 cycle per minute

Exclusion Criteria:

* Minors
* Pregnant or lactating women
* Patient without social security
* Patient hospitalize without consent
* Chest pain with acute coronary electro-cardiographic change leading immediate achievement of a diagnostic coronary angiography and/or therapeutic
* Pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency and unit intensive care patient.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ARA SOMOHANO Claire, PH, Principal Investigator — Emergency NGO Onlus
Locations (1):
- University Hospital Grenoble, Grenoble, Grenoble, France